CLINICAL TRIAL: NCT02484599
Title: Evaluation of a Computerized Attention Training (CAT) to Modify Attention Bias for Food Cues in Anorexia Nervosa Patients
Brief Title: Look at Food and Lose Your Fear - Evaluation of a Computerized Attention Training (CAT) for Anorexia Nervosa Patients
Acronym: CAT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS ID 160749
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Anorexia Nervosa
Keywords: Eating Disorders; Anorexia Nervosa; Attention bias; Attention bias modification
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAT active attention bias modification (Experimental): Active computerized attention training (CAT). Attention training via repeated trials of a modified anti-saccade task with concurrent assessment of eye-movements intended to direct attention towards food stimuli using pictorial food and non-food stimuli (see Werthmann, Field, Roefs, Nederkoorn, & Jansen, 2014).
  Interventions: Behavioral: Computerized attention training (CAT)
- CAT sham bias modification (Placebo Comparator): Sham computerized attention training. Attention training via repeated trials of a modified anti-saccade task with concurrent assessment of eye-movements not intended to change attention processing of food stimuli using pictures of two different non-food stimuli categories (e.g. household and musical instruments).
  Interventions: Behavioral: Sham computerized attention training (control condition)

INTERVENTIONS:
Behavioral: Computerized attention training (CAT) — Three sessions of active computerized attention training.
  Other Names: Attention bias modification training
  Arms: CAT active attention bias modification
Behavioral: Sham computerized attention training (control condition) — Three sessions of sham computerized attention training.
  Arms: CAT sham bias modification

SUMMARY:
The purpose of this study is to test the therapeutic effects of a computerized attention training for patients with Anorexia Nervosa (AN). The primary aim is to determine if a computerized attention training can modify attention towards food and ameliorate eating disorder symptoms and related difficulties, such as anxiety. The secondary aim is to explore underlying mechanisms that contribute to these improvements. The stability of potentially observed effects over a one-month period will also be determined.

DETAILED DESCRIPTION:
Recently, attention bias modification (ABM) has successfully been applied in the field of anxiety disorders and emerging evidence suggests that attention bias modification can ameliorate attention bias for threatening stimuli. ABM is based on the premise that if biased attention maintains disorder symptoms, a modification of the bias should reduce symptoms. The advantage of ABM is that it operates implicitly, thereby offering a more indirect, less deliberate procedure. This requires less cognitive control compared to the effortful and explicit psychotherapeutic treatment of cognitive biases. As food-related fears and avoidance in AN patients have been recognized as important anxiety-related symptoms, ABM seems particularly suitable to treat food-related fears and avoidance, especially because AN patients might be unaware of their avoidance strategy. The aim of this study is to test if food-related fears and food avoidance can be changed by experimentally modifying attention towards food in Anorexia Nervosa patients using an innovative computerized training paradigm (computerized attention training - CAT) and to evaluate related change in symptoms.

The investigators hypothesize that the active CAT will change attentional processing of food cues (research aim 1), transfer to changes in food-related fears and food avoidance, and to improvements in AN symptoms and weight in the short term (research aim 2) and longer term (research aim 3).

ELIGIBILITY:
Inclusion Criteria:

* BMI < 18.5 5 kg/m2
* Current diagnosis of AN-restricting type, AN-Binge/purging type or Eating Disorder Not Otherwise Specified (EDNOS) - Anorexia type
* Fluent in English

Exclusion Criteria:

* Currently taking a dose of any psychoactive medication that has not been stable for at least 14 days prior to participation in the study
* Currently meeting the diagnostic criteria of another major psychiatric disorder (e.g., major depressive disorder, substance dependence, schizophrenia or bipolar disorder) needing treatment in its own right
* Learning and developmental impairments
* If the disorder is currently life threatening
* If patients are currently suicidal
* If patients are currently having extreme physiological complications or co-morbid alcohol and drug-abuse disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-10 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Attention bias | max. 2 weeks (pre and post attention bias modification training)
  The dot-probe task with concurrent assessment of eye-movements will be used for the assessment of attention bias at baseline and post-treatment.

SECONDARY OUTCOMES:
Eating Disorder symptoms | max. 2 week (pre and post attention bias modification training) and at 4 weeks follow-up
  The Eating Disorder Examination Questionnaire (EDE-Q, Fairburn & Belgin, 1994) is a commonly used index for AN symptoms and will be assessed at baseline and post-treatment and at 4 weeks follow-up.
Body Mass Index | max. 2 (pre and post attention bias modification training) and after 4 weeks (follow-up).
  Weight and height will be assessed to calculate BMI and assess whether BMI changes occurred during the study period due to CAT

OTHER OUTCOMES:
Eating Behaviour | max. 2 weeks
  Participants will be instructed to taste from different food options and their willingness to do so and their actual intake will be assessed as measure for behavioural food avoidance at baseline and at post-treatment.
Approach and avoidance tendencies | max. 2 weeks
  Approach and avoidance tendencies for food pictures will be assessed with the Affective Simon Task (AST, see Neimeijer, de Jong, & Roefs, 2015) at baseline and at post-training to test changes in food-related approach or avoidance.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Werthmann, PhD, Principal Investigator — Institute of Psychiatry, Psychology and Neuroscience, King's College London
Locations (1):
- Institute of Psychiatry, Psychology and Neuroscience, London, United Kingdom

REFERENCES:
- [Background] Neimeijer RA, de Jong PJ, Roefs A. Automatic approach/avoidance tendencies towards food and the course of anorexia nervosa. Appetite. 2015 Aug;91:28-34. doi: 10.1016/j.appet.2015.03.018. Epub 2015 Mar 24. PMID 25817483
- [Background] Werthmann J, Field M, Roefs A, Nederkoorn C, Jansen A. Attention bias for chocolate increases chocolate consumption--an attention bias modification study. J Behav Ther Exp Psychiatry. 2014 Mar;45(1):136-43. doi: 10.1016/j.jbtep.2013.09.009. Epub 2013 Sep 29. PMID 24140811